CLINICAL TRIAL: NCT01807208
Title: PLATFORM to Maximize Patient Knowledge of Health Goals After Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00034650; 5U19HS021092 (AHRQ)
Record Dates: First submitted 2013-02-28; First posted 2013-03-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2016-02

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute myocardial infarction; patient education; prevention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational tool (Experimental): Patients randomized to the educational tool arm of the study will receive mailed educational materials at 1 week post hospital discharge and again at 3 months after discharge.
  Interventions: Other: Educational Tool
- Usual care (No Intervention): Patients in this arm of the study will receive usual care.

INTERVENTIONS:
Other: Educational Tool — A personalized health goal education and reminder tool, with 3 parts: "report card" showing the status of secondary prevention domains during hospitalization; questions to help prepare the patient for the follow-up visit; and potential questions for the physician.
  Arms: Educational tool

SUMMARY:
The goals of this study are two fold: 1) To learn whether a personalized patient health goal and reminder tool helps patients to learn more about their condition and to make changes in behavior and medication taking to reduce the risk of another heart attack. 2) To examine a blood sample to learn how patients are responding to their medications. The study team will enroll approximately 220 patients in the hospital recovering from a heart attack. Half of the patients will receive the educational tools and a copy will be sent to their outpatient provider.

DETAILED DESCRIPTION:
The goals of this study are two fold: 1) To evaluate the impact of a personalized patient health goal education and reminder tool on patient adherence to evidence based therapies and subsequent cardiovascular risk factor modification after acute myocardial infarction (AMI); 2) To assess age-related heterogeneity in antiplatelet response among AMI patients. This is a prospective study of ~220 AMI patients, with at least half over age 65 years. Patients will be surveyed with questionnaires (at baseline and 6 months post discharge) and biomarkers (baseline only) to assess the status of their physical function, depression, nutrition, inflammation, and response to antiplatelet therapies. Patients will also be administered a walking test and a grip strength test at baseline. About 1 week after hospital discharge, and again about 3 months after hospital discharge, about half of the patients and their outpatient providers will receive the personalized post-AMI health goal education and reminder tool on patient adherence to evidence-based secondary prevention therapies. Data will be analyzed in aggregate using descriptive statistics. The primary endpoint of interest is a composite measure of adherence at six months to secondary prevention therapies described as the sum of measures received divided by the sum of available opportunities. The secondary endpoint will be analyzed to describe platelet response profiles as a function of age. The study team anticipates the risks for this study to be minimal, since the patient does not receive any investigational therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with either ST-elevation MI (STEMI) or non-ST-elevation MI (NSTEMI) who are on antiplatelet therapy at the time of enrollment.
2. English language literacy and
3. Able to provide written informed consent.

Exclusion Criteria:

1. Patients less than 18 years of age.
2. Patients who are unable or unwilling to comply with the protocol or not expected to complete the study period, including its follow-up requirements
3. Life expectancy less than 6 months or discharged on hospice care.
4. Patients without at least 1 scheduled outpatient follow-up visit inside the Duke University Affiliated Physicians network.
5. Patients who receive a coronary artery bypass grafting (CABG) during the eligible enrollment hospitalization.
6. Active chronic inflammatory conditions (e.g., inflammatory bowel disease, lupus, rheumatoid arthritis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2013-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in the effect of patient health goal and reminder tool on health outcomes | baseline, 6 months
  The study team plans to evaluate the impact of a personalized patient health goal education and reminder tool on 6-month clinical and other health outcomes. The measure will be a composite of lab measures (such as blood pressure at goal; BMI at goal), behavior change (physical activity, smoking cessation) and medication use (beta blockers, angiotensin-converting enzyme inhibitors (ACEI)/ angiotensin receptor blockers (ARBs), statins if not contraindicated)
Satisfaction and usefulness of education tools | 6 months
  The study team will ask patients whether they used the education tools in their follow-up physician visits post-AMI; how helpful the tools were; whether they were easy to read and understand; and whether the amount of material presented was appropriate

SECONDARY OUTCOMES:
Age-associated changes that modulate antiplatelet response | index hospitalization (average 3-5 days), 6 months post discharge
  Describe the physical and functional changes (inflammation, functional decline, nutrition and depression) that modulate platelet inhibitory response to anti-platelet medications
Association between antiplatelet response and subsequent bleeding events | 6 months
  Explore the association between antiplatelet response and subsequent bleeding events (number and location of bleeds) among AMI patients to optimize risk stratification and individualize treatment using clinical, physical function and laboratory data
Age-associated variation in platelet inhibitory response | index hospitalization (average 3-5 days)
  To examine blood biomarkers of platelet inhibitory response and variability in these biomarkers between younger (less than or equal to 70 years of age) and older patients (over 70 years)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Peterson, MD, MPH, Study Chair — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No